CLINICAL TRIAL: NCT03503669
Title: Reducing Risk for Alzheimer's Disease in High-Risk Women Through Yogic Meditation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Alzheimer's Research and Prevention Foundation (Other)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-001876
Record Dates: First submitted 2018-04-11; First posted 2018-04-20 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Memory impairment; Meditation; Yoga; Memory Training; Mild Cognitive Impairment; MCI; Geriatric; fMRI; Alzheimer's disease; Cardiovascular risk
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Memory Disorders | interventions — Cognitive Training; Meditation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memory Training (Active Comparator): Group memory training will be administered for amnestic mild cognitive impairment (MCI)
  Interventions: Behavioral: Memory Training
- Kundalini yoga and meditation (Experimental): Participants will engage in weekly yoga classes and daily 12 minute meditation
  Interventions: Behavioral: Kundalini yoga and meditation

INTERVENTIONS:
Behavioral: Memory Training — Participants will attend a weekly memory training class for 12 weeks as well as receive daily memory homework (12 minute duration) for the 12 weeks.
  Arms: Memory Training
Behavioral: Kundalini yoga and meditation — Participants will participate in a 60 minute yoga and meditation session weekly for 12 weeks and will be assigned a daily Kirtan Kriya meditation (12 minute duration) for 12 weeks.
  Arms: Kundalini yoga and meditation

SUMMARY:
The purpose of this pilot study will be to test whether Kundalini yoga (KY) and Kirtan Kriya (KK) yogic meditation is superior to Memory Enhancement Training (MET) for improving cognitive functioning, health (including cardiovascular factors), and mood in women with high AD risk.

DETAILED DESCRIPTION:
Overall, the investigators anticipate recruiting 100 women (50 or older) with MCI and high Alzheimer's disease risk. Subjects will either receive: (1) MET class for 60 minutes per week; or (2) Kundalini yoga and "Kirtan Kriya" meditation class for 60 minutes per week. Assessments will be completed immediately after the interventions at 6 and 12 weeks and follow-up visits at week 24 and 48 to monitor the overall benefit of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Amnestic MCI, as defined by a Clinical Dementia Rating Scale score of .5.
2. High cardiovascular risk defined as at least one of the following:

   * 7.5 percentile risk or higher using ASCVD risk calculator
   * Myocardial Infarction more than 6 months ago
   * Diabetes
   * Taking medication for blood pressure > 140/90 blood pressure
   * Taking medication for lyperlipidemia LDL >160
3. Sufficient English proficiency and the 8th grade or higher reading level as determined by the word reading subtest of the Wide Range Achievement Test-IV (this criterion is necessary in order to ensure ability to participate in MET, which involves reading and writing and has a Flesch-Kinkaid school equivalency of 7th grade)
4. Capacity to provide informed consent

Exclusion Criteria:

1. History of psychosis, bipolar disorder, alcohol/ drug dependence, or neurological disorder
2. Recent (within three months) surgery, anticipated surgery within next year, or unstable medical condition
3. Any disability preventing participation in MET or KK+KY (e.g., severe visual or hearing impairment)
4. Insufficient English proficiency to participate in either MET or KK+KY
5. Diagnosis of dementia
6. Mini Mental Health Examination score of 23 or below
7. Currently taking any psychoactive medication
8. Participation in a psychotherapy that involves cognitive training
9. Practice of Kundalini Yoga or Kirtan Kriya within the past year
10. Myocardial Infarction within the past 6 months

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, MS, MD, Principal Investigator — UCLA Semel Institute
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krause-Sorio B, Siddarth P, Kilpatrick L, Milillo MM, Aguilar-Faustino Y, Ercoli L, Narr KL, Khalsa DS, Lavretsky H. Yoga Prevents Gray Matter Atrophy in Women at Risk for Alzheimer's Disease: A Randomized Controlled Trial. J Alzheimers Dis. 2022;87(2):569-581. doi: 10.3233/JAD-215563. PMID 35275541
- [Derived] Grzenda A, Siddarth P, Milillo MM, Aguilar-Faustino Y, Khalsa DS, Lavretsky H. Cognitive and immunological effects of yoga compared to memory training in older women at risk for alzheimer's disease. Transl Psychiatry. 2024 Feb 14;14(1):96. doi: 10.1038/s41398-024-02807-0. PMID 38355715
- [Derived] Kilpatrick LA, Siddarth P, Krause-Sorio B, Milillo MM, Aguilar-Faustino Y, Ercoli L, Narr KL, Khalsa DS, Lavretsky H. Impact of Yoga Versus Memory Enhancement Training on Hippocampal Connectivity in Older Women at Risk for Alzheimer's Disease. J Alzheimers Dis. 2023;95(1):149-159. doi: 10.3233/JAD-221159. PMID 37482992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 100 participants were consented and completed screen visit while 79 participants completed baseline and were randomized to either group. 10 individuals were screen fails and 11 dropped out before randomization.
Period: Overall Study
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Started | 39 | 40
Completed | 37 | 26
Not Completed | 2 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memory Training | Kundalini Yoga and Meditation | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.3) | 65.5 (9.1) | 66.48 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 36 | 33 | 69
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 27 | 32 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79
Hopkins Verbal Learning Test (HVLT) [Mean (Standard Deviation); unit: units on a scale] — Hopkins Verbal Learning Test (HVLT) is a verbal memory task with 12 words learned over three trials, with the correct words summed for the Total Recall score (range = 0 - 36), with higher scores representing better performance.
  units on a scale | 26.66 (5.48) | 28.02 (5.29) | 27.34 (5.40)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hopkins Verbal Learning Test (HVLT) Total Recall Score
Description: Verbal memory was measured with the Hopkins Verbal Learning Test (HVLT) total recall scores. The HVLT form contains 12 nouns, four words each from one of three semantic categories (e.g., precious gems, articles of clothing, vegetables, etc.), to be learned over the course of three learning trials. When scoring the HVLT, the three learning trials are combined to calculate a total recall score. Total scores range from 0-36 with higher scores indicating better outcome.
Time Frame: Measured at Baseline and Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Number analyzed (Participants) | 37 | 26
units on a scale | -0.94 (5.10) | -1.65 (6.90)
Statistical Analysis 1: Comparison: Memory Training vs Kundalini Yoga and Meditation; Test type: Superiority; p > 0.05, Mixed Models Analysis

2. Primary Outcome: Change in Delayed Recall Cognitive Domain Scores
Description: Delayed Recall Cognitive Domain score was constructed from: HVLT Delayed Recall, Rey-Osterrieth Complex Figure Test [30-minute Delayed Recall], WMS-IV Logical Memory II Delayed Recall.
  Raw scores were transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. A z-score of 0 represents the sample mean. These z-scores were then averaged to produce a Delayed Recall Cognitive Domain score. Higher Delayed Recall Cognitive Domain scores are indicative of better performance.
Time Frame: Measured at Baseline and Week 24
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Number analyzed (Participants) | 37 | 26
z-score | 0.02 (0.55) | -0.31 (0.37)
Statistical Analysis 1: Comparison: Memory Training vs Kundalini Yoga and Meditation; Test type: Superiority; p = 0.008, Mixed Models Analysis

3. Primary Outcome: Change in Executive Function Cognitive Domain Scores
Description: Executive Function Cognitive Domain score was constructed from:
  Trail Making Test A and B, Stroop Interference [Golden version] and FAS.
  Raw scores were transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. A z-score of 0 represents the sample mean. These z-scores were then averaged to produce an Executive Function Cognitive Domain score. Higher Executive Function Cognitive Domain scores are indicative of better performance.
Time Frame: Measured at Baseline and Week 24
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Number analyzed (Participants) | 37 | 26
z-score | -0.03 (0.70) | -0.04 (0.42)
Statistical Analysis 1: Comparison: Memory Training vs Kundalini Yoga and Meditation; Test type: Superiority; p > 0.05, Mixed Models Analysis

4. Secondary Outcome: Change in Memory Functioning Questionnaire (MFQ) Scale
Description: Secondary outcome measures included the Memory Functioning Questionnaire (MFQ), a self-assessment scale. The MFQ is a scale that assesses subjective memory complaints. We will use the following MFQ subscales: General Frequency of Forgetting (MFQ factor 1), Seriousness of Forgetting (MFQ factor 2), and Retrospective Functions (MSQ factor 3). Each item is scored from 1 to 7 with higher scores indicating a higher level of perceived memory functioning. MSQ factor 1 (33 items) ranges from 7 to 231, MFQ factor 2 (18 items) ranges from 7-126 and MSQ factor 3 (5 items) ranges from 7 to 35.
Time Frame: Measured at Baseline and Week 24, change from baseline to week 24 is reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Number analyzed (Participants) | 37 | 26
units on a scale
  MFQ Factor 1 | 0.29 (0.75) | 0.54 (1.03)
  MFQ Factor 2 | -0.30 (1.34) | 0.64 (1.24)
  MFQ Factor 3 | 0.51 (1.58) | 0.70 (1.04)
Statistical Analysis 1: Comparison: Memory Training vs Kundalini Yoga and Meditation; Test type: Superiority; p > 0.05, Mixed Models Analysis

5. Secondary Outcome: Change in Medical Outcomes Study Short Form 36-Item Health Survey (SF-36)
Description: Health-Related quality of life will be determined using the Medical Outcomes Study Short Form 36-Item Health Survey (SF-36) which comprises 8 scales: physical functioning, role limitations - physical, role limitations - emotional, energy, emotional well-being, social functioning, pain, and general health. Scales are scored from 0 to 100 with higher scores indicating higher quality of life.
Time Frame: Measured at Baseline and Week 24, change from baseline to week 24 is reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Number analyzed (Participants) | 37 | 26
units on a scale
  Physical Functioning | 0.60 (26.47) | 2.70 (20.48)
  Role Physical | -15.90 (40.41) | 3.12 (39.91)
  Role Emotional | -18.18 (44.16) | 2.77 (46.01)
  Energy | -2.42 (18.96) | 0.83 (18.80)
  Emotional Wellbeing | 0.72 (14.01) | -3.33 (19.00)
  Social Functioning | 0 (24.60) | -9.89 (36.29)
  Pain | -4.92 (17.35) | -7.50 (25.31)
  General Health | 1.06 (13.33) | -1.45 (16.18)
Statistical Analysis 1: Comparison: Memory Training vs Kundalini Yoga and Meditation; Test type: Superiority; p > 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline through study completion, up to six months.
Description: Adverse events were assessed by asking participants whether they experienced any negative side effects
Arm/Group | Memory Training | Kundalini Yoga and Meditation
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 3/39 | 3/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memory Training (N=39) | Kundalini Yoga and Meditation (N=40)
Food Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Vaccine side effect (Immune system disorders) | 0 (0) | 1 (1)
Flu (Immune system disorders) | 0 (0) | 1 (1)
COVID-19 (Immune system disorders) | 1 (1) | 0 (0)
Steroid Injection (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
After March 18th, 2020, all assessments were completed remotely due to COVID-19 until restrictions were lifted for eligible participants to come in-person.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03503669/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT03503669/ICF_001.pdf